CLINICAL TRIAL: NCT04375709
Title: Health-related Quality of Life (HRQOL) and Physical Performance in Individuals After COVID-19 Induced Hospitalisation and the Impact of a Standard Care Follow-up Program: a Longitudinal Observational Cohort Study
Brief Title: Quality of Life and Physical Performance After Novel Coronavirus Infection (COVID-19);
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_00899 / COV19_2020
Record Dates: First submitted 2020-05-04; First posted 2020-05-05 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Covid-19 (New Coronavirus) Infection
Keywords: COVID-19; SARS-V2; Quality of Life; Physical Performance
MeSH Terms: conditions — COVID-19; Infections | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Physical exercise — The intervention consists out of combined aerobic and strength exercise supervised and guided by specialized physical therapists; additional methods like functional electrical stimulation or oxygen supplementation are added during the main training if indicated.
Behavioral: Education sessions — Sessions include information on physical activity (behaviour), coping with stress and anxiety, dyspnoe, or fatigue; Professional support is given in case of risk for nutritional deficits or post-traumatic stress; sessions are conducted by medical specialists or specialized physiotherapists. All sessions are individually-tailored. In case of nutrition or psychological issues individual sessions are guided by specific health-professionals.

SUMMARY:
This study aims to observe the long-term health-related quality of life (HRQOL) and physical performance in individuals hospitalized due to a COVID-19 infection. Therefore, data is extracted from a study-site standard aftercare program which has been adjusted for this patient population. This comprehensive aftercare program includes education sessions and physical exercise. A second aim is to observe adherence and feasibility to the program and if indicated compare the clinical data and outcomes from patients following the program with patients denying to participate in guided exercise and education sessions.

It is expected that patients hospitalized due to COVID-19 infection show a reduction in physical performance and HRQOL directly after discharge. The severity of illness is hypothesized to be associated with a reduction as well in HRQOL and physical performance after one-year post-discharge.

DETAILED DESCRIPTION:
Currently, the U.S. National Library of Medicine (April 2nd) reports 282 studies registered investigating the COVID-19 infection. According to the present knowledge the COVID-19, also known as novel type Coronavirus or SARS-CoV-2 (severe acute respiratory syndrome-Coronavirus-2), belongs to a large family of viruses consist-ing of hundreds of variations and subtypes of this virus (World Health Organisation (WHO)/emergencies, April 2nd 2020). These types of virus' can cause respiratory and gastrointestinal symptoms ranging from a mild cold to pneumonia. The clinical manifestation of this novel type of Coronavirus - COVID-19 - was found to cause more severe pneumonia or severe acute respiratory syndrome such as the acute respiratory distress syndrome (ARDS). According to the data of Arabi and colleagues (2020) average age in Chinese affected individuals were 60, 40% had comorbid conditions, 42% required invasive mechanical ventilation and the mortality rate was at 62%. Epidemiological information from other countries is not yet published. According to the WHO in the Europe Region, 503730 cases and 33617 deaths were reported since January 25th 2020. In the 8,5 million populated countries of Switzerland, the number of confirmed cases raised to 23'574 and 756 deaths (Bundesamt für Gesundheit) Situationsbericht, April 9th). According to this report, the incidence of infection and hospitalization is highest in individuals aged 50 and older with a higher presence registered in men. Nevertheless, a certain number of affected individuals is between 20 and 50 years which is in accordance with the number presented from large studies in China (50.7%-55.1%). Among the 23'674 positive tested 2730 are currently hospitalized. Among these 280 individuals require mechanically assisted ventilation, meaning health care at an intensive care unit (status April 2nd).

In this acute situation of the pandemic, there is an enormous urge to finding a vaccine or medications to release or prevent severe symptoms and complications due to the new virus. Therefore, in the listed studies keen interest is on drug interventions to stop the expansion of this virus. However, knowledge on long-term consequences of physical condition and psychological state is unknown. Although, taking into account the clinical manifestation observed in the severe cases negative long-term consequences have to be expected as described in the following paragraph.

Up to date knowledge exist on the clinical manifestation which varies from asymptomatic to severe disease with approximately 80% of the cases found to present an asymptomatic carrier.

Thus, about 13.8% to 35% is suffering a severe course including dyspnoea, respiratory frequency ≥30/minute, desaturation of blood oxygen (≤93%) and or lung infiltrates >50% of the lung within 24-48 hours. Further signs of hospitalized individuals are fever, cough, myalgia, fatigue and sputum production. In literature, the clinical picture is described as bilateral pneumonia or acute respiratory distress syndrome which leads to a severe organ failure of the lung. These patients require oxygen therapy with invasive (17%) or non-invasive (14%) mechanically assisted ventilation. And the higher probability of preloaded organ dysfunctions due to co-morbidities most often high blood pressure (13%), diabetes (4-6%) and COPD (1-5%) has to be taken into account.

According to the WHO report and Lai et al (2020) between 6.1% to 28%, respectively, were found to be in a critical stage. Acute respiratory failure, septic shock and/ or multiple organ failure defined this stage. According to a retrospective analysis from a large population in Wuhan, these patients require intensive care with most of them presenting (multi) organ failure with acute respiratory distress (ARDS, 67%), acute kidney injury (29%), cardiac injury (23%), and liver dysfunction (29%). These patients require invasive or non-invasive mechanical ventilation. The mortality rate for critically ill COVID-19 patients varies from 1-4% to 4.3% according to large studies reported by Lai et al. (2020).

According to these statistics, about 4.3% of the 280 patients requiring intensive care in Switzerland (n=12) would not survive. Taking the current number of 2730 hospitalised patients reported above, these statistics result in about 2718 individuals surviving severe illness in Switzerland. A critical point is the high risk of the length of stay on the ward as explained in the following paragraph.

Patients in the severe and critical state are likely to suffer prolonged length of stay in the hospital according to Lia et al. (2020) and Wang et al. (2020) (±21 days). Studies on ARDS and critically ill patients led to strong evidence that prolonged length of stay, particularly with prolonged mechanical ventilation, leads to a significant negative impact on lung function, physical activity and emotional state. For example, from 109 patients suffered an ARDS (age interquartile from 35 to 57) the 5 years follow up showed a relevant reduction on physical condition (76% of the distance in the 6 Minute Walk Test (6MWT)) when compared to age and sex-matched norm values. Interestingly, these deficits were found despite normal to "near"-normal pulmonary function. A recent post-hoc analysis on 116 patients mechanically ventilated for at least >24h showed that a longer duration of mechanical ventilation and exposure to norepinephrine were associated with intensive-care-unit acquired weakness (ICU-AW; defined as <48/100 on the Medical Research Council Score). Hatch et al. (2018) for example found in their multicenter follow-up study, that 46% of the survivors of critical illness suffered from anxiety, 40% from depression and 22% from post-traumatic stress disorder (PTSD). In the specific population of ARDS survivors (n=74) numbers are slightly lower ranging from moderate to severe depression in 16% and 23%, respectively and for anxiety 24% and 23% at 1 and 2 years, respectively. These findings on survivors of ARDS and critical illness underline the assumption that survivors of a COVID-19 induced hospitalized will suffer from physical and psychological long-term consequences.

In research on critical illness post-ICU, only moderate evidence and large risk of bias exist on the effect of follow-up rehabilitation post-ICU. However, some qualitative studies support the thought that patients might need additional care after discharge home. King et al. (2019) investigated in their scoping review of qualitative studies the needs of critical illness survivors and found that after discharge home patients had continuing information needs on understanding their critical illness and coping with the long-term sequelae and stress.

These qualitative findings were underlined and supported by quantitative studies investigating long-term effects in this population. In patients who suffered an acute respiratory failure greatest change in physical function was found two months after discharge. And in ICU survivors requiring one or more weeks of mechanical ventilation the degree of disability one week after ICU discharge was predictive for physical and mental recovery and mortality in the one-year follow up.

In contrast to the findings on critical illness aftercare programs were found having a positive impact in a population with pulmonary disease. In survivors of ARDS due to severe influenza, A pneumonitis an 8-week pulmonary rehabilitation program improved significantly exercise capacity and quality of life improved significantly. And in patients with chronic obstructive pulmonary disease (COPD), the American Thoracic Society recommends respiratory rehabilitation early after discharge. Furthermore, according to the NICE guidelines "Rehabilitation after critical illness in adults" patients with rehabilitation needs should be seen two to three months after hospital discharge and should be reassessed to establish health and social care needs.

Additionally, based on an expert consensus following questions are still unanswered and considered as being relevant for the rehabilitation of these patients. Some examples are listed below:

* "What proportion of COVID-19 survivors have (extra-pulmonary) physical, functional, emotional and sociable treatable traits, justifying rehabilitation…?"
* "What types of patients will exist post-COVID-19 (e.g. good recovery, frailty, persistent respiratory impairment) and in what proportion?"
* "What is the impact of a COVID-19-related prolonged ward stay on physical and emotional functioning?
* What are the opportunities to intervene early, immediately post-acute hospital discharge?
* For how long after hospital discharge are COVID-19 survivors contagious? The latter two questions are cardinal to provide safe and feasible rehabilitation post-acute hospital discharge. To present the feasibility and safety of the aftercare program developed and conducted on the study site a short excurse on literature is provided.

Recent knowledge (published February 28 and 1st of April) from high impact journals give following solid time frames on viral shedding according to the traceability of Covid-19 RNA. Reverse transcription-polymerase chain reaction (RT-PCR) of virus RNA was used to measure the quantity of virus RNA in both studies.

Wölfel and colleagues isolated the virus daily from sputum, pharyngeal swabs, and stool since the first day of symptom onset. The samples were taken from individuals with mild to moderate symptoms (e.g. symptoms of lung affection). Maximal viral load was found before 5 days in these participants with the mild course being highest in stool and sputum. Based on their findings authors state that being 10 days beyond symptoms and less than 100,000 viral RNA copies per ml of sputum do have a little residual risk of infectivity, based on cell culture. Ling et al., isolated viral RNA from 66 participants post-Covid-19 infection as well from the stool, urine, and blood specimens during the convalescence. These samples were obtained from patients who survived a severe course of infection. The longest duration from onset of symptoms to first negative RT-PCR results for oropharyngeal swabs of convalescent patients was 22 days.

Zhou et al. (2020) studied as well the viral shedding with the daily analysis using PCR of Covid-19 throat swab specimens from 191 patients. For survivors, the duration of viral shedding showed an interquartile range of 17 to 22 days in patients with severe disease status (survivors). In summary, current knowledge shows the duration of viral traceability and thus the risk of infection from 10 to 22 days in patients with mild and severe illness, respectively. The average time to incubation found ranged from 5.2 to 12.5 days (Zhou et al., 2020) and average hospital duration ranged from 7 to 15 days in the 425 patients from Wuhan.

Therefore, subtracting lowest period of incubation (5 days) from the maximal duration of viral shedding (22 days) resulting in 17 days after first confirmed diagnose to be safe for hospital on-site testing. Based on this data and adding the criteria 4 days without specific COVID-19 symptoms (described in chapter 6.2.1), the committee developing the specific aftercare program - from which data will be taken for this study - considered as safe and feasible inviting patients post-acute hospital discharge when 14 days post diagnose and the mentioned four days (total ≥18 days).

In summary, there is a lack of knowledge on long term consequences of physical, emotional and quality of life outcomes. The similarity of clinical manifestation of the COVID-19 infection with ARDS or/and critical illness leads to the consideration of evidence found in this patient population. This evidence points out the high risk of long-term deficits on the above-mentioned outcomes and the relevance of patient-tailored rehabilitation programs.

Therefore, we consider it as essential to gather and analyse data on short and long-term quality of life and physical performance of patients after hospitalization due to COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at the Kantonsspital Winterthur (KSW) due to COVID-19 infection (laboratory-confirmed),

  * with or without mechanically assisted ventilation
  * being at risk to obtain severe illness caused by the COVID-19*
  * individuals without defined risk factors but requiring oxygenation during hospitalisation
* Agree to general consent or specific consent to subsequent use of his/her personal health data for research purpose
* German-speaking

Exclusion Criteria:

* Presence of mental disability or impairments to reasoning or judgment
* Individuals who are immunocompromised due to medical treatment
* A documented objection of subsequent use of personal health data

Specific exclusion criteria for presence at the hospital (for evaluation and training); criteria will be verified during the phone-based screening process. After two weeks of a COVID-19 positive diagnosis and with four entire days the patient reports no signs of:

* fever >37.3° C
* sore throat,
* cough (productive or non-productive)
* common cold

Also, treatment-based immunocompromised patients are excluded for on-site evaluation and training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult individuals after COVID-19 infection hospitalized at the Kantonsspital Winterthur (Switzerland)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life; EuroQoL (EQ-5D-5L) | 01.04.2020 - 30.05.2021
  Self-managed questionnaire on functional status, anxiety, pain and independence in daily living; The EuroQoL includes a five item scale and a visual analog scale from 0-100 in order to quantify perception of current health.
  The five item scale includes ordinary scores from 0-5. Lower numbers equal less problems and better quality of life.
  For the visual analog scale a higher number represents a better health status perceived.
6-minute walk test | 01.04.2020 - 30.05.2021
  6-minute walk test measures the distance acquired during six minutes walking, it quantifies the physical performance, dyspnoea and endurance.

SECONDARY OUTCOMES:
Jamar dynamometer | 01.04.2020 - 30.05.2021
  Measures the handgrip strength and is associated with sarcopenia, mortality and independence in life (e.g. for older individuals and patients after or with critical illness)
Hospital Anxiety and Depression Scale (HADS) | 01.04.2020 - 30.05.2021
  Self-administered questionnaire on anxiety and depression after hospitalization; bot, anxiety and depression is quantified by an ordinal scale from 0-3, respectively. The lower the number the less signs of depression or anxiety are present.
revised Impact of Event Scale (IES-R) | 01.04.2020 - 30.05.2020
  Questionnaire on avoidance, intrusion and arousal (or overreaction) in order to identify potential risk for post-traumatic stress. The Scale includes 22 questions ordinally scored from "not at all" to " very frequent" with four scores. The scores are transformed into numbers (0,1,3,5). The values are put in a formula resulting in a single value.A value below zero indicates no risk of post-traumatic stress disorder (PTSD) is present. Values equal or higher than zero indicate the risk of a PTSD
Mini-Nutritional Assessment (MNA) | 01.04.2020 - 30.05.2021
  Questionnaire on the nutritional condition of the patient. It includes 16 questions and 2 measures. Points range from 0-30; A score <17 indicates malnutirtion, a score from 17-23.5 indicates a risk of malnutrition and scores between 24-30 indicate normal nutritional behaviour.
Spirometry (bed-side) | 01.04.2020 - 30.05.2021
  Measures the lung function (bedside screening)
Post-Covid Functional Scale (PCFS) | 01.04.2020 - 30.05.2021
  This scale measures the functional state and Independence of patients after COVID-19 infection. The scale includes two items scored from 0-4 and 0-5. A high value indicates more restrictions in function and independence during daily life.
modified Medical Research Council Dyspnoea Scale (mMRC Dyspnoea) | 01.04.2020 - 30.05.2021
  Quantifies and stratifies the perception of dyspnoea with a score ranging from 0-4. The higher the value the more frequent and more severe is the perception of dyspnoea during daily life activities.

CONTACTS AND LOCATIONS:
Overall Officials: David Gisi, Study Director — Kantonsspital Winterthur KSW; Martina Betschart, PhD, Principal Investigator — Kantonsspital Winterthur KSW; Spencer Rezek, MSc Cand., Study Chair — Kantonsspital Winterthur KSW; Ines Unger, MSc Cand., Study Chair — Kantonsspital Winterthur KSW; Natalie Ott, MSc Cand., Study Chair — Kantonsspital Winterthur KSW; Swantje Beyer, MD, Study Chair — Kantonsspital Winterthur KSW; Markus Hofer, MD, Study Chair — Kantonsspital Winterthur KSW; Karrer Urs, PD MD, Study Chair — Kantonsspital Winterthur KSW; Giuseppe Mungo, MSc, Study Chair — Kantonsspital Winterthur KSW; Cornel Sieber, Prof. MD, Study Director — Kantonsspital Winterthur KSW
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arabi YM, Murthy S, Webb S. Correction to: COVID-19: a novel coronavirus and a novel challenge for critical care. Intensive Care Med. 2020 May;46(5):1087-1088. doi: 10.1007/s00134-020-06009-2. PMID 32189010
- [Background] Bohannon RW. Muscle strength: clinical and prognostic value of hand-grip dynamometry. Curr Opin Clin Nutr Metab Care. 2015 Sep;18(5):465-70. doi: 10.1097/MCO.0000000000000202. PMID 26147527
- [Background] Dres M, Jung B, Molinari N, Manna F, Dube BP, Chanques G, Similowski T, Jaber S, Demoule A. Respective contribution of intensive care unit-acquired limb muscle and severe diaphragm weakness on weaning outcome and mortality: a post hoc analysis of two cohorts. Crit Care. 2019 Nov 21;23(1):370. doi: 10.1186/s13054-019-2650-z. PMID 31752937
- [Background] Gandotra S, Lovato J, Case D, Bakhru RN, Gibbs K, Berry M, Files DC, Morris PE. Physical Function Trajectories in Survivors of Acute Respiratory Failure. Ann Am Thorac Soc. 2019 Apr;16(4):471-477. doi: 10.1513/AnnalsATS.201806-375OC. PMID 30571923
- [Background] Hatch R, Young D, Barber V, Griffiths J, Harrison DA, Watkinson P. Anxiety, Depression and Post Traumatic Stress Disorder after critical illness: a UK-wide prospective cohort study. Crit Care. 2018 Nov 23;22(1):310. doi: 10.1186/s13054-018-2223-6. PMID 30466485
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Hosey MM, Bienvenu OJ, Dinglas VD, Turnbull AE, Parker AM, Hopkins RO, Neufeld KJ, Needham DM. The IES-R remains a core outcome measure for PTSD in critical illness survivorship research. Crit Care. 2019 Nov 19;23(1):362. doi: 10.1186/s13054-019-2630-3. No abstract available. PMID 31744551
- [Background] Hsieh MJ, Lee WC, Cho HY, Wu MF, Hu HC, Kao KC, Chen NH, Tsai YH, Huang CC. Recovery of pulmonary functions, exercise capacity, and quality of life after pulmonary rehabilitation in survivors of ARDS due to severe influenza A (H1N1) pneumonitis. Influenza Other Respir Viruses. 2018 Sep;12(5):643-648. doi: 10.1111/irv.12566. Epub 2018 Jun 12. PMID 29676537
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] King J, O'Neill B, Ramsay P, Linden MA, Darweish Medniuk A, Outtrim J, Blackwood B. Identifying patients' support needs following critical illness: a scoping review of the qualitative literature. Crit Care. 2019 May 24;23(1):187. doi: 10.1186/s13054-019-2441-6. PMID 31126335
- [Background] Lai CC, Liu YH, Wang CY, Wang YH, Hsueh SC, Yen MY, Ko WC, Hsueh PR. Asymptomatic carrier state, acute respiratory disease, and pneumonia due to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2): Facts and myths. J Microbiol Immunol Infect. 2020 Jun;53(3):404-412. doi: 10.1016/j.jmii.2020.02.012. Epub 2020 Mar 4. PMID 32173241
- [Background] Ling Y, Xu SB, Lin YX, Tian D, Zhu ZQ, Dai FH, Wu F, Song ZG, Huang W, Chen J, Hu BJ, Wang S, Mao EQ, Zhu L, Zhang WH, Lu HZ. Persistence and clearance of viral RNA in 2019 novel coronavirus disease rehabilitation patients. Chin Med J (Engl). 2020 May 5;133(9):1039-1043. doi: 10.1097/CM9.0000000000000774. PMID 32118639
- [Background] Major ME, Kwakman R, Kho ME, Connolly B, McWilliams D, Denehy L, Hanekom S, Patman S, Gosselink R, Jones C, Nollet F, Needham DM, Engelbert RH, van der Schaaf M. Surviving critical illness: what is next? An expert consensus statement on physical rehabilitation after hospital discharge. Crit Care. 2016 Oct 29;20(1):354. doi: 10.1186/s13054-016-1508-x. PMID 27793165
- [Background] Sillen MJ, Franssen FM, Delbressine JM, Vaes AW, Wouters EF, Spruit MA. Efficacy of lower-limb muscle training modalities in severely dyspnoeic individuals with COPD and quadriceps muscle weakness: results from the DICES trial. Thorax. 2014 Jun;69(6):525-31. doi: 10.1136/thoraxjnl-2013-204388. Epub 2014 Jan 7. PMID 24399630
- [Background] Singh SJ, Puhan MA, Andrianopoulos V, Hernandes NA, Mitchell KE, Hill CJ, Lee AL, Camillo CA, Troosters T, Spruit MA, Carlin BW, Wanger J, Pepin V, Saey D, Pitta F, Kaminsky DA, McCormack MC, MacIntyre N, Culver BH, Sciurba FC, Revill SM, Delafosse V, Holland AE. An official systematic review of the European Respiratory Society/American Thoracic Society: measurement properties of field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1447-78. doi: 10.1183/09031936.00150414. Epub 2014 Oct 30. PMID 25359356
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Taito S, Yamauchi K, Tsujimoto Y, Banno M, Tsujimoto H, Kataoka Y. Does enhanced physical rehabilitation following intensive care unit discharge improve outcomes in patients who received mechanical ventilation? A systematic review and meta-analysis. BMJ Open. 2019 Jun 9;9(6):e026075. doi: 10.1136/bmjopen-2018-026075. PMID 31182443
- [Background] Tipping CJ, Young PJ, Romero L, Saxena MK, Dulhunty J, Hodgson CL. A systematic review of measurements of physical function in critically ill adults. Crit Care Resusc. 2012 Dec;14(4):302-11. PMID 23230880
- [Background] Wolfel R, Corman VM, Guggemos W, Seilmaier M, Zange S, Muller MA, Niemeyer D, Jones TC, Vollmar P, Rothe C, Hoelscher M, Bleicker T, Brunink S, Schneider J, Ehmann R, Zwirglmaier K, Drosten C, Wendtner C. Virological assessment of hospitalized patients with COVID-2019. Nature. 2020 May;581(7809):465-469. doi: 10.1038/s41586-020-2196-x. Epub 2020 Apr 1. PMID 32235945
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Zanini A, Aiello M, Adamo D, Casale S, Cherubino F, Della Patrona S, Raimondi E, Zampogna E, Chetta A, Spanevello A. Estimation of minimal clinically important difference in EQ-5D visual analog scale score after pulmonary rehabilitation in subjects with COPD. Respir Care. 2015 Jan;60(1):88-95. doi: 10.4187/respcare.03272. Epub 2014 Oct 21. PMID 25336531
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- See also: Verified the 27th of April — https://srs-mcmaster.ca/wp-content/uploads/2020/04/Rehabilitation-for-Patients-with-COVID-19-Apr-08-2020.pdf
- See also: verified the 2nd of April 2020 — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/events-as-they-happen
- See also: verified the 2nd of April 2020 — https://who.maps.arcgis.com/home/item.html?id=9bc9d986ff5a4c6c850682873a94da47
- See also: verified the 9nd of April 2020 — https://www.who.int/publications-detail/report-of-the-who-china-joint-mission-on-coronavirus-disease-2019-(covid-19)
- See also: Guidelines on management of critical illness; verified the 9th of April 2020 — https://www.nice.org.uk/guidance/qs158/resources/rehabilitation-after-critical-illness-in-adults-pdf-75545546693317